CLINICAL TRIAL: NCT00544752
Title: Indoor Temperature and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Ass Prof Karl Franklin, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 03-563; NCT01315600 (obsolete NCT alias)
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea syndromes, ambient indoor temperature
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 16 (Experimental): indoor temperature of 16 degrees celcius
  Interventions: Other: 16
- 20 (Experimental): indoor temperature 20 degrees celcius
  Interventions: Other: indoor temperature of 20 degrees celcius
- 24 (Experimental): indoor temperature of 24 degrees celcius
  Interventions: Other: indoor temperature of 24 degrees celcius

INTERVENTIONS:
Other: 16 — indoor temperature of 16 degrees celcius
  Arms: 16
Other: indoor temperature of 20 degrees celcius — indoor temperature of 20 degrees celcius
  Arms: 20
Other: indoor temperature of 24 degrees celcius — indoor temperature of 24 degrees celcius
  Arms: 24

SUMMARY:
The purpose of this study is to test whether different indoor temperature affect the frequency of sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea

Exclusion Criteria:

* Central sleep apnea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index, karolinska sleepiness scale | one night

SECONDARY OUTCOMES:
Sleep stages, sleep efficiency | One night

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, PhD, Principal Investigator — Dept Respiratory Medicine, University Hospital, Umeå
Locations (1):
- Dept of respiratory medicine, Umeå, Sweden

REFERENCES:
- [Derived] Valham F, Sahlin C, Stenlund H, Franklin KA. Ambient temperature and obstructive sleep apnea: effects on sleep, sleep apnea, and morning alertness. Sleep. 2012 Apr 1;35(4):513-7. doi: 10.5665/sleep.1736. PMID 22467989